CLINICAL TRIAL: NCT01549938
Title: Cholecalciferol Intervention to Prevent Respiratory Infections Study: a Double-blind Randomised Controlled Trial to Evaluate the Efficacy of 20,000 IU/wk Cholecalciferol in Reducing Respiratory Tract Infection in a Cohort of Healthy Young Adults
Brief Title: Cholecalciferol Intervention to Prevent Respiratory Infections Study
Acronym: CIPRIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menzies Institute for Medical Research (Other)
Collaborators: Royal Hobart Hospital Research Foundation (funding source) (Unknown)
Responsible Party: Principal Investigator, Dr Steve Simpson, Jr., Postdoctoral Research Associate, Menzies Institute for Medical Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIPRIS; ACTRN12612000054819 (Registry Identifier: Australia and New Zealand Clinical Trials Registry); U1111-1126-9425 (Registry Identifier: World Health Organisation Universal Trial Number)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Respiratory Tract Infection; Vitamin D Deficiency
Keywords: Vitamin D; Cholecalciferol; Respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): 20,000 IU cholecalciferol capsule
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator): Microcellulose capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 20,000 IU cholecalciferol capsule, given once weekly for 16 weeks.
  Arms: Treatment
Dietary Supplement: Placebo — Microcellulose capsule identical in appearance to treatment
  Arms: Placebo

SUMMARY:
This is a feasibility double-blind randomised controlled trial in 32 participants. It evaluates the feasibility of a full trial which will examine the efficacy of weekly supplementation of cholecalciferol (vitamin D3) relative to placebo on the subsequent frequency and severity of objectively-verified symptomatic acute respiratory tract infection, overall and as a proportion of detected colonisations of the upper respiratory tract by 9 of the most common aetiologic viral pathogens.

DETAILED DESCRIPTION:
The hypotheses of the full study are:

Primary The group treated with vitamin D3 will have a significantly lower frequency of symptomatic respiratory tract infections than controls.

Secondary

1. Among persons with detected viral colonisations of the nasopharynx, treated persons will have a lower frequency of symptomatic respiratory tract infection resultant than controls.
2. Treated group will have significantly less severe symptomatic RTIs than controls.
3. Treated group will have significantly shorter symptomatic RTI durations than controls.

For the pilot, a cohort of 32 healthy young adults satisfying inclusion criteria will be randomised to cholecalciferol supplement or identical placebo and evaluated daily for the occurrence of RTI symptoms and evaluated weekly for the presence of respiratory colonisation by relevant pathogens using nasopharyngeal swab and polymerase chain reaction using selected pathogen-specific primers. This pilot will demonstrate the logistic feasibility of the proposed study design and provide preliminary data which will inform a larger study to be undertaken next year.

ELIGIBILITY:
Inclusion Criteria:

* Students undertaking study at the MS1 building of University of Tasmania Medical Sciences Precinct (17 Liverpool St Hobart TAS) for the full duration between May and September 2012

Exclusion Criteria:

* Persons who have used tobacco within the 6 months preceding study entry
* Persons who have used any vitamin D (cholecalciferol or ergocalciferol) supplements or calcium supplements within the 3 months preceding study entry and/or persons who refuse to not start taking any such supplement during the study
* Persons using any immunomodulatory medication, diuretic medication, antiepileptic medication, or barbiturates.
* Persons who presently have been diagnosed with any chronic infectious disease (e.g. HIV, tuberculosis), chronic immune deficiency or autoimmune condition, or respiratory condition (e.g. asthma, chronic obstructive pulmonary disease).
* Persons who are hypersensitive to vitamin D.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Frequency of validated respiratory tract infections during study period | 17 weeks
  Frequency of validated respiratory tract infections during study period. Acute respiratory tract infections defined by respiratory symptoms reported by daily online survey lasting over a day and verified at exam by study nurse.

SECONDARY OUTCOMES:
Proportion of colonisations leading to symptomatic respiratory tract infections | 17 weeks
  Proportion of colonisations with respiratory pathogens that go on to symptomatic verified respiratory tract infections. Colonisation detected by nasal swab sampled quantitiative RT-PCR.
Severity of respiratory tract infections during study | 17 weeks
  Severity (objective and subjective) of respiratory tract infections during the study. Subjective severity of symptoms reported by Likert scale (0-5) for each symptom. Objective severity by number and duration of symptoms.
Mean duration of respiratory tract infections during study | 17 weeks
  Mean duration of respiratory tract infections during study. Duration defined as number of days from participant-reported symptom onset to sympton resolution, as reported in daily online questionnaire.
Frequency of non-respiratory tract infections during study | 17 weeks
  Frequency of non-respiratory tract infections during study. Non-respiratory tract infections defined by non-respiratory symptoms reported by daily online survey lasting over a day and verified at exam by study nurse.
Concentration of serum 25-hydroxyvitamin D by the end of the study | 17 weeks
  Concentration of serum 25-hydroxyvitamin D by the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Steve Simpson, Jr., PhD, MPH, Principal Investigator — Menzies Institute for Medical Research
Locations (1):
- Menzies Research Institute Tasmania, Hobart, Tasmania, Australia